CLINICAL TRIAL: NCT06698770
Title: Leveraging Behavioral Science to Improve Medicine Optimization Conversations With Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of Sydney (Other)
Responsible Party: Principal Investigator, Vordenberg, Clinical Associate Professor of Clinical Pharmacy and Associate Chair, Clinical Pharmacy, College of Pharmacy, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: HUM00259517
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2024-11

CONDITIONS: Deprescribing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Start medication - Lower chance of future health problems (Experimental): Participants read a hypothetical scenario where a doctor recommends starting a new medication to lower their chances of experiencing significant health problems.
  Interventions: Other: Anticipated long-term use of medication; Other: Period re-evaluation of medication
- Start medication - Higher risk without medication (Experimental): Participants read a hypothetical scenario where a doctor recommends starting a new medication because they could experience a higher risk of serious health problems without it
  Interventions: Other: Anticipated long-term use of medication; Other: Period re-evaluation of medication
- Stop medication - Lack of benefit (Experimental): Participants read a hypothetical scenario where a doctor suggests stopping the medication due to a lack of benefit.
  Interventions: Other: Anticipated long-term use of medication; Other: Period re-evaluation of medication
- Stop medication - Potential for harm (Experimental): Participants read a hypothetical scenario where a doctor suggests stopping the medication due to the potential for harm.
  Interventions: Other: Anticipated long-term use of medication; Other: Period re-evaluation of medication

INTERVENTIONS:
Other: Anticipated long-term use of medication — In this hypothetical scenario, the doctor anticipates that the participant will take this medication for the rest of their life.
Other: Period re-evaluation of medication — In this hypothetical scenario, the doctor anticipates that the participant will take this medication for the rest of their life but will periodically re-evaluate the benefits and risks of the medication.

SUMMARY:
Our online, survey-based experiment will include 2,400 adults who are 65-years and older (n=1,200 each from United States and Australia). Each participant will be asked to give their opinions on a hypothetical patient scenario that has been developed by our diverse team in partnership with our stakeholder organizations.This work is expected to significantly contribute to our understanding of how older adults make decisions about deprescribing medications.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older and resides in Australia or the United States

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 2420 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Preference regarding starting medication | 1 year
  Response to statement, "Based on what you have read so far, what would you prefer to do with this diabetes medicine?" on a 6-point Likert scale with scale anchors 1=Strongly prefer not to start medicine and 6=Strongly prefer to start medicine
Stopping medication | 1 year
  Response to statement, "Based on what you have read so far, what would you prefer to do with this diabetes medicine?" on a 6-point Likert scale with scale anchors 1=Strongly prefer not to continue and 6=Strongly prefer to stop

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No